CLINICAL TRIAL: NCT03169933
Title: Combined, Intensified and Modulated Adjuvant Therapy in Prostate Carcinoma: a Phase II Trial
Brief Title: Combined, Intensified and Modulated Adjuvant Therapy in Prostate Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Howard University (Other); University of Bologna (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIMA-1
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: adjuvant; androgen suppressive therapy; literature review; phase II; prostate neoplasms; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intensified and modulated adjuvant RT (Other): All patients underwent combined, intensified and modulated adjuvant radiotherapy for 5 days a week with the following doses: 1) pelvic node irradiation (45 Gy; 1.8 Gy/fraction) followed by boost on the prostate bed (19.8-25.2 Gy; 1.8 Gy/fraction; total dose: 64.8-70.2 Gy) or 2) exclusive prostate bed irradiation (64.8 -70.2 Gy; 1.8 Gy/fraction).
  Interventions: Radiation: Combined, intensified and modulated adjuvant radiotherapy

INTERVENTIONS:
Radiation: Combined, intensified and modulated adjuvant radiotherapy
  Other Names: adjuvant androgen deprivation therapy

SUMMARY:
Patients with high risk prostate cancer may benefit from radiotherapy after radical prostatectomy. The investigators postulated that adjuvant androgen deprivation therapy (ADT), radiation dose escalation, and selective pelvic irradiation may improve outcome. A phase II trial was designed to prove that combined-intensified-modulated-adjuvant (CIMA) treatment may improve 5-year biochemical relapse free survival (bRFS) from 75% to 90% in high risk patients. The delivered dose to tumor bed and pelvic nodes was 64.8-70.2 Gy and 45 Gy (57% of patients), respectively, and 69% received ADT.

DETAILED DESCRIPTION:
Prostate cancer patients at high risk of loco-regional recurrences may benefit from postoperative radiotherapy (RT) following radical prostatectomy (EORTC trial 22911). However, despite an improvement in biochemical relapse-free survival (bRFS), the risk of recurrences remained high for those patients. The investigators postulated that adjuvant androgen deprivation therapy (ADT), radiation dose escalation, and selective pelvic irradiation for patients at risk for regional failures may improve the outcome. The combined-intensified-modulated-adjuvant (CIMA) as described may improve survival through a reduction of loco-regional and systemic failures.

A phase II trial was designed to test the hypothesis that CIMA treatment may improve 5-year bRFS by 15%. Patients less than 80 years old, with a histological diagnosis of prostate adenocarcinoma without distant metastases, stage pT2-4 N0-1, no previous treatments and an ECOG performance status of 0-2 were selected. All patients had at least one of these pathologic features: extracapsular extension, positive surgical margins, or seminal vesicle invasion. Radiation dose to the tumor bed ranged from 64.8 to 70.2 Gy. Pelvic lymph nodes were treated to 45 Gy in selected patients at risk of regional failures (57%). Selected patients at risk for distant metastases (69.1%) received hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* < 80 years old
* histological diagnosis of prostate adenocarcinoma
* no distant metastases
* stage pT2-4
* N0-1
* ECOG performance status of 0-2
* One of these pathologic features: extracapsular extension, positive surgical margins, or seminal vesicle invasion. extracapsular extension, positive surgical margins or seminal vesicle invasion, or positive lymph-nodes
* No surgical complications such as pelvic infections or lymphocele, intraoperative rectal injury or severe urinary incontinence
* Preoperative and postoperative PSA test, bone scan and CT-scan or MRI of abdomen and pelvis prior to enrolment
* Normal bone marrow function

Exclusion Criteria:

* Previously treated with Radiotherapy
* Previously treated with androgen deprivation therapy
* Previously treated with chemotherapy for prostate cancer. They also had to be free

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2004-01-02 (Actual); Primary Completion 2009-01-10 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Biochemical relapse free survival | Five years
  Survival free from increase of PSA level exceeding 0.2 ng/mL for those with postsurgical PSA level of 0.2 ng/mL or lower, and as two consecutive PSA increases for patients with a postsurgical PSA level of > 0.2 ng/ml

SECONDARY OUTCOMES:
Incidence of early treatment-emergent adverse events | < 90 days.
  Adverse events after radiotherapy . Acute side effects were scored according to the Radiation Therapy Oncology Group (RTOG) scale.
Incidence of late treatment-emergent adverse events were assessed with Radiation Morbidity Scoring Scheme of the RTOG/European Organization for Research and Treatment of Cancer (EORT) | 5 years
  Late complications were assessed with the Late Radiation Morbidity Scoring Scheme of the RTOG/European Organization for Research and Treatment of Cancer (EORT)
First evidence of any pelvic recurrence | 5 years
  First evidence of any pelvic recurrence
Metastasis-free survival | 5 years
  The first evidence of any extra pelvic recurrence of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Study Director — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mantini G, Siepe G, Alitto AR, Buwenge M, Nguyen NP, Farioli A, Schiavina R, Catucci F, Deodato F, Fionda B, Frascino V, Macchia G, Ntreta M, Padula GDA, Arcelli A, Cammelli S, Rambaldi GZ, Cilla S, Valentini V, Morganti AG. Tailored postoperative treatment of prostate cancer: final results of a phase I/II trial. Prostate Cancer Prostatic Dis. 2018 Nov;21(4):564-572. doi: 10.1038/s41391-018-0064-7. Epub 2018 Jul 23. PMID 30038390